CLINICAL TRIAL: NCT07295522
Title: Pharmacological Optimization in Prevention in Heart Failure: A Sex-gap?
Acronym: PopS-HF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Massimo Piepoli, Professor, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PopS-HF; 2025-520660-18 (EudraCT Number)
Record Dates: First submitted 2025-12-01; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Acute Heart Failure; Heart Failure With Reduced Ejection Fraction (HFrEF); Heart Failure With Preserved Ejection Fraction (HFPEF); Heart Failure With Mildly Reduced Ejection Fraction
Keywords: heart failure; women; GDMT; Pharmacological Optimization; phase IV; High intensity up-titration; Secondary prevention; Sex differences; Real world data
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: A parallel-group design is used, with participants randomized 1:1 to receive either high-intensity optimization of guideline-directed medical therapy or usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Participants in the usual care arm will receive sequential introduction and adjustment of guideline-directed medical therapy (GDMT) according to the treating cardiologist or general physician's clinical judgment, following routine practice. Follow-up will occur at weeks 6, 12, 24, 36, and 52 after randomization, with clinical visits and intermediate phone contacts as per standard care.
- High-intensity care (Experimental): Participants assigned to the high-intensity arm will begin rapid initiation and optimization of guideline-directed medical therapy (GDMT) according to the STRONG-HF protocol. During hospitalization, eligible therapies (beta-blockers (BB), Angiotensin converting enzyme inhibitor(ACEi) /Angiotensin II receptor blocker (ARB)/Angiotensin Receptor-Neprilysin Inhibitors(ARNI), Mineralocorticoid Receptor Antagonists (MRA), and Sodium-Glucose Co-Transporter inhibitor 2 (SGLT2i) for HFrEF/HFmrEF; MRA and SGLT2i for HFpEF will be prescribed at least at half of the recommended target dose. Further titration toward full optimal doses will be performed within the first 6 weeks if clinically appropriate. Participants will undergo clinical assessments at weeks 2, 4, 6, 12, 24, 36, and 52, with safety monitoring including vital signs, physical examination, and laboratory evaluation (NT-proBNP, electrolytes, kidney function). Additional visits may occur after any up-titration if needed for safety.
  Interventions: Drug: Guideline-Directed Medical Therapy (GDMT)

INTERVENTIONS:
Drug: Guideline-Directed Medical Therapy (GDMT) — Guideline-directed medical therapy (GDMT) including beta-blockers, ACE inhibitors or ARBs or ARNIs, mineralocorticoid receptor antagonists, and SGLT2 inhibitors, all approved and commercially available, used according to current ESC guidelines.
  Participants in the high-intensity care arm are assigned to a strategy of rapid initiation and optimization of GDMT based on the STRONG-HF protocol. Eligible therapies (beta-blockers, ACEi/ARB/ARNI, mineralocorticoid receptor antagonists, and SGLT2 inhibitors for HFrEF/HFmrEF; MRA and SGLT2 inhibitors for HFpEF) are started during hospitalization at least at half of the recommended target dose, followed by frequent clinical assessments and dose titration, when clinically appropriate, within 6 weeks. Safety monitoring includes clinical examination, vital signs, laboratory tests (NT-proBNP, electrolytes, kidney function), and additional visits after each titration if needed.
  Arms: High-intensity care

SUMMARY:
The goal of this clinical trial is to learn whether a rapid and intensive optimization of heart failure medications in women can improve outcomes after hospitalization for heart failure. It will also investigate the safety and the tolerance of these treatments when given at full guideline-recommended doses.

The main questions it aims to answer are:

1. Does intensive medication optimization reduce death or hospital readmissions for heart failure within one year?
2. Do women benefit as much as men from intensive and full-dose heart failure therapy?
3. Is this treatment protocol safe and feasible also in women?

Researchers will compare two groups of women hospitalized for heart failure:

* High-intensity care: starting and increasing all recommended heart-failure medications as quickly as possible and monitoring patients closely during the first weeks after discharge.
* Usual care: medications are started and adjusted gradually, according to the judgment of the treating cardiologist and the patient's usual care team.

The study will follow participants for 12 months to see whether the high-intensity strategy reduces death, hospital readmission for heart failure, or worsening symptoms. It will also evaluate side effects, medication tolerance, and quality of life.

Participants will be randomly assigned to one of the two groups, attend regular follow-up visits for one year, complete a short quality-of-life questionnaire (EQ-5D).

This study will include about 360 women from 13 hospitals in Italy. It is sponsored by IRCCS Policlinico San Donato and funded by the Italian Medicines Agency (AIFA).

DETAILED DESCRIPTION:
PopS-HF is a phase IV, low-interventional, multicenter randomized controlled trial designed to test whether intensive optimization of guideline directed medical therapy (GDMT), following the STRONG-HF (Safety, Tolerability and Efficacy of Rapid Optimization, Helped by NT-proBNP Testing of Heart Failure Therapies) titration strategy, improves outcomes in women hospitalized for heart failure (HF).

The study also includes a retrospective analysis of national healthcare databases and specialized HF registries from 2018-2023 to evaluate how GDMT are prescribed in real-world practice and to identify sex-related differences in treatment patterns and outcomes.

Eligible patients are women aged 18-85 years hospitalized for acute HF with evidence of congestion and hemodynamic stability before discharge. Exclusion criteria include severe comorbidities, pregnancy, and inability to follow up.

The prospective component randomizes 368 patients to an intensive strategy or usual care, with follow-up visits at 2, 4, 6, 12, 24, 36, and 52 weeks.

The primary endpoint is a composite of all-cause mortality, HF readmission, or worsening HF within 1 year.

Secondary endpoints assess optimization of therapy, side effects, biomarkers (NT-proBNP), and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients >18 <85 years.
2. Hospital admission within the 72 hours prior to Screening for acute heart failure with dyspnea at rest and pulmonary congestion on chest X-ray, and other signs and/or symptoms of heart failure such as edema and/or positive rales on auscultation.
3. All measures within 24 hours prior to Randomization of systolic blood pressure ≥ 100 mmHg, and of heart rate ≥ 60 bpm.
4. All measures within 24 hours prior to Randomization of serum potassium ≤ 5.0 mEq/L (mmol/L).
5. Biomarker criteria for persistent congestion:

   5.1. At Screening, NT-proBNP >1,800 pg/mL (2,350 pg/mL in case of atrial fibrillation) 5.2. At the time of Randomization (1-2 days prior to discharge), NT-proBNP >1,000 pg/mL (1,300 pg/mL in case of Atrial Fibrillation) to ensure the persistence of congestion and the acuity of the index episode).
6. At 1 week prior to admission, at Screening, and at Visit 2 6.1. If EF<50% (ie HFrEF or HFmrEF) either <½ the optimal dose of ACEi/ARB/ARNi and MRA and BB or no SGLT2i (see Table) must have been prescribed 6.2. If EF>50% (ie HFpEF): <½ the optimal dose of MRA (see Table) or no SGLT2i.
7. Written informed consent to participate in the study.

Exclusion Criteria:

1. Male patients
2. Age < 18 or > 85 years.
3. Mechanical ventilation (not including CPAP/BIPAP) in the 24 hours prior to Screening.
4. Significant pulmonary disease contributing substantially to the patients' dyspnoea such as FEV1 <1 liter or need for chronic systemic or nonsystemic steroid therapy, or any kind of primary right heart failure such as primary pulmonary hypertension or recurrent pulmonary embolism.
5. Myocardial infarction, unstable angina or cardiac surgery within 3 months, or cardiac resynchronization therapy (CRT) device implantation within 3 months, or percutaneous transluminal coronary intervention (PTCI), within 1 month prior to Screening or during the index event.
6. Index Event (admission for Acute Heart Failure) triggered primarily by a correctable aetiology such as significant arrhythmia (e.g., sustained ventricular tachycardia, or atrial fibrillation/flutter with sustained ventricular response >130 beats per minute, or bradycardia with sustained ventricular arrhythmia <45 beats per minute), infection, severe anaemia, acute coronary syndrome, pulmonary embolism, exacerbation of Chronic Obstructive Pulmonary Disease (COPD), planned admission for device implantation or severe non-adherence leading to very significant fluid accumulation prior to admission and brisk diuresis after admission. Troponin elevations without other evidence of an acute coronary syndrome are not an exclusion.
7. Uncorrected thyroid disease, active myocarditis, or known amyloid or hypertrophic obstructive cardiomyopathy.
8. History of heart transplant or on a transplant list or using or planned to be implanted with a ventricular assist device.
9. Sustained ventricular arrhythmia with syncopal episodes within the 3 months prior to screening that is untreated.
10. Presence at Screening of any hemodynamically significant valvular stenosis or regurgitation, except mitral or tricuspid regurgitation secondary to left ventricular dilatation, or the presence of any hemodynamically significant obstructive lesion
11. Active infection at any time during the AHF hospitalization prior to Randomization based on abnormal temperature and elevated WBC or need for intravenous antibiotics.
12. Stroke or Transient Ischemic Attack (TIA) within the 3 months prior to Screening.
13. Primary liver disease considered to be life threatening.
14. Renal disease or eGFR < 30 mL/min/1.73m2 (as estimated by the simplified MDRD formula) at Screening or history of dialysis.
15. Psychiatric or neurological disorder, cirrhosis, or active malignancy leading to a life expectancy < 6 months.
16. Prior (defined as less than 30 days from screening) or current enrollment in a CHF trial or participation in an investigational drug or device study within the 30 days prior to screening or 5 half-lives of the study drug, whichever is longer.
17. Discharge for the AHF hospitalization anticipated to be >14 days from admission, or to a long-term care facility. Randomization must occur within 12 days following admission and at 1-2 days prior to anticipated discharge.
18. Inability to comply with all study requirements, due to major co-morbidities, social or financial issues or a history of noncompliance with medical regimens, that might compromise the patient's ability to understand and/or comply with the protocol instructions or follow-up procedures.
19. Pregnant or nursing (lactating) women.
20. Hypersensitivity to the active substance or to any of the excipients as indicated in Summary of Product Characteristics of Investigational Medicinal Product (IMPs).
21. Angioedema.
22. Severe heart failure (NYHA class IV).

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2027-06-08 (Estimated); Study Completion 2028-06-08 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality, heart failure (HF) readmission, or worsening HF within 1 year. | 12 months
  Composite endpoint including occurrence of (1) death from any cause, (2) hospital readmission for heart failure, or (3) clinically assessed worsening of heart failure.

SECONDARY OUTCOMES:
Optimization of Beta-blocker Therapy | 12 months
  Percentage of participants achieving dose optimization of beta-blockers according to guideline-recommended targets or maximum tolerated dose.
Optimization of ACEi/ARB/ARNI Therapy | 12 months
  Proportion of participants achieving dose optimization of ACE inhibitors, angiotensin receptor blockers, or angiotensin receptor-neprilysin inhibitors according to guideline-recommended targets or maximum tolerated dose.
Optimization of Mineralocorticoid Receptor Antagonists (MRAs) | 12 months
  percentage of participants achieving dose optimization of MRAs at recommended dose or maximum tolerated dose.
Optimization of SGLT2 Inhibitors | 12 months
  Percentage of poulation achieving full implementation of SGLT2 inhibitors
Discontinuation of GDMT due to side effects | 12 months
  Percentage of participants discontinuing any GDMT class (beta-blockers, ACEi/ARB/ARNI for EF <50%, MRAs, or SGLT2 inhibitors) due to adverse effects or intolerance.
NT-proBNP Changes | 12 months
  Change in plasma NT-proBNP levels from baseline to follow-up visits in each study arm.
Quality of Life (EQ-5D-5L Score) | 12 months
  Change in health-related quality of life measured by the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire. The EQ-5D-5L also includes a visual analogue scale (VAS) ranging from 0 to 100, with higher scores indicating better perceived health status.
One-year All-Cause Mortality | 12 months
  Incidence of death from any cause within 12 months after randomization.
One-year Heart Failure Readmission | 12 months
  Incidence of hospital readmission for heart failure within 12 months after randomization.
One-year Worsening Heart Failure | 12 months
  Incidence of worsening heart failure within 12 months after randomization, defined as deterioration of heart failure signs and symptoms requiring urgent escalation of therapy, including emergency department visit or outpatient intravenous diuretic therapy.

OTHER OUTCOMES:
Exploratory Subgroup Analyses | 12 months
  Evaluation of treatment effects across predefined subgroups, including EF <50% vs ≥50%, age <65 vs ≥65 years, diabetes, chronic kidney disease, obesity.

CONTACTS AND LOCATIONS:
Locations (13):
- Italy (13):
  - IRCCS Policlinico San Donato, San Donato Milanese, MILANO
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - Azienda Sanitaria Locale Bari, Bari
  - Azienda USL Toscana Nord Ovest - Cecina, Cecina
  - Ospedale Universitario di Ferrara, Ferrara
  - Azienda USL Toscana Centro, Florence
  - Centro Cardiologico Monzino, Milan
  - Istituto Auxologico Italiano, Milan
  - Fondazione Toscana Gabriele Monasterio, Pisa
  - Ospedale S. Maria delle Croci, Ravenna
  - Azienda USL IRCCS Di Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Universitario Campus Bio-medico, Roma
  - Ospedale San Camillo Forlanini, Roma

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will not be made publicly available. Data sharing is restricted due to ethical and regulatory requirements under GDPR and Italian data protection regulations. Aggregate study results will be published.

REFERENCES:
- [Background] Okumura N, Jhund PS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Swedberg K, Zile MR, Solomon SD, Packer M, McMurray JJ; PARADIGM-HF Investigators and Committees*. Importance of Clinical Worsening of Heart Failure Treated in the Outpatient Setting: Evidence From the Prospective Comparison of ARNI With ACEI to Determine Impact on Global Mortality and Morbidity in Heart Failure Trial (PARADIGM-HF). Circulation. 2016 Jun 7;133(23):2254-62. doi: 10.1161/CIRCULATIONAHA.115.020729. Epub 2016 Apr 20. PMID 27143684
- [Background] Brotons C, Falces C, Alegre J, Ballarin E, Casanovas J, Cata T, Martinez M, Moral I, Ortiz J, Perez E, Rayo E, Recio J, Roig E, Vidal X. Randomized clinical trial of the effectiveness of a home-based intervention in patients with heart failure: the IC-DOM study. Rev Esp Cardiol. 2009 Apr;62(4):400-8. doi: 10.1016/s1885-5857(09)71667-6. English, Spanish. PMID 19401125
- [Background] Mebazaa A, Davison B, Chioncel O, Cohen-Solal A, Diaz R, Filippatos G, Metra M, Ponikowski P, Sliwa K, Voors AA, Edwards C, Novosadova M, Takagi K, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G. Safety, tolerability and efficacy of up-titration of guideline-directed medical therapies for acute heart failure (STRONG-HF): a multinational, open-label, randomised, trial. Lancet. 2022 Dec 3;400(10367):1938-1952. doi: 10.1016/S0140-6736(22)02076-1. Epub 2022 Nov 7. PMID 36356631
- [Background] Dewan P, Rorth R, Jhund PS, Shen L, Raparelli V, Petrie MC, Abraham WT, Desai AS, Dickstein K, Kober L, Mogensen UM, Packer M, Rouleau JL, Solomon SD, Swedberg K, Zile MR, McMurray JJV. Differential Impact of Heart Failure With Reduced Ejection Fraction on Men and Women. J Am Coll Cardiol. 2019 Jan 8;73(1):29-40. doi: 10.1016/j.jacc.2018.09.081. PMID 30621948
- [Background] Lainscak M, Milinkovic I, Polovina M, Crespo-Leiro MG, Lund LH, Anker SD, Laroche C, Ferrari R, Coats AJS, McDonagh T, Filippatos G, Maggioni AP, Piepoli MF, Rosano GMC, Ruschitzka F, Simic D, Asanin M, Eicher JC, Yilmaz MB, Seferovic PM; European Society of Cardiology Heart Failure Long-Term Registry Investigators Group. Sex- and age-related differences in the management and outcomes of chronic heart failure: an analysis of patients from the ESC HFA EORP Heart Failure Long-Term Registry. Eur J Heart Fail. 2020 Jan;22(1):92-102. doi: 10.1002/ejhf.1645. Epub 2019 Dec 20. PMID 31863522
- [Background] Butler J, Yang M, Sawhney B, Chakladar S, Yang L, Djatche LM. Treatment patterns and clinical outcomes among patients <65 years with a worsening heart failure event. Eur J Heart Fail. 2021 Aug;23(8):1334-1342. doi: 10.1002/ejhf.2252. Epub 2021 Jun 17. PMID 34053163
- [Background] Fiuzat M, Ezekowitz J, Alemayehu W, Westerhout CM, Sbolli M, Cani D, Whellan DJ, Ahmad T, Adams K, Pina IL, Patel CB, Anstrom KJ, Cooper LS, Mark D, Leifer ES, Felker GM, Januzzi JL, O'Connor CM. Assessment of Limitations to Optimization of Guideline-Directed Medical Therapy in Heart Failure From the GUIDE-IT Trial: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2020 Jul 1;5(7):757-764. doi: 10.1001/jamacardio.2020.0640. PMID 32319999
- [Background] Kapelios CJ, Murrow JR, Nuhrenberg TG, Montoro Lopez MN. Effect of mineralocorticoid receptor antagonists on cardiac function in patients with heart failure and preserved ejection fraction: a systematic review and meta-analysis of randomized controlled trials. Heart Fail Rev. 2019 May;24(3):367-377. doi: 10.1007/s10741-018-9758-0. PMID 30618017
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Najafi F, Jamrozik K, Dobson AJ. Understanding the 'epidemic of heart failure': a systematic review of trends in determinants of heart failure. Eur J Heart Fail. 2009 May;11(5):472-9. doi: 10.1093/eurjhf/hfp029. Epub 2009 Feb 27. PMID 19251729
- [Background] Piepoli MF, Adamo M, Barison A, Bestetti RB, Biegus J, Bohm M, Butler J, Carapetis J, Ceconi C, Chioncel O, Coats A, Crespo-Leiro MG, de Simone G, Drexel H, Emdin M, Farmakis D, Halle M, Heymans S, Jaarsma T, Jankowska E, Lainscak M, Lam CSP, Lochen ML, Lopatin Y, Maggioni A, Matrone B, Metra M, Noonan K, Pina I, Prescott E, Rosano G, Seferovic PM, Sliwa K, Stewart S, Uijl A, Vaartjes I, Vermeulen R, Verschuren WM, Volterrani M, Von Haehling S, Hoes A. Preventing heart failure: a position paper of the Heart Failure Association in collaboration with the European Association of Preventive Cardiology. Eur J Prev Cardiol. 2022 Feb 19;29(1):275-300. doi: 10.1093/eurjpc/zwab147. PMID 35083485
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992